CLINICAL TRIAL: NCT02167178
Title: Investigation of the Relationship Between Oesophageal Doppler Assessed Increases in Cardiac Output and Microvascular Visceral Blood Flow in Healthy Volunteers
Brief Title: The Relationship Between Cardiac Output and Microvascular Visceral Blood Flow
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: A12012012
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Saline Solution; Sodium Chloride; contrast agent BR1

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Volunteers receiving 0.9% NaCl: Volunteers receiving 0.9% NaCl to optimise stroke volume
  Interventions: Other: Administration of 0.9% NaCl solution; Other: Measurement of stroke volume; Other: Measurement of microvascular blood flow
- Volunteers receiving gelofusine: Volunteers receiving gelofusine to optimise stroke volume
  Interventions: Other: Measurement of stroke volume; Other: Measurement of microvascular blood flow; Other: Administration of gelofusine

INTERVENTIONS:
Other: Administration of 0.9% NaCl solution — Volunteers administered 0.9% NaCl solution in 250ml boluses
  Other Names: Normal saline; Saline
  Groups: Volunteers receiving 0.9% NaCl
Other: Measurement of stroke volume — The measurement of stroke volume will be performed using an Oesophageal Doppler Monitor.
Other: Measurement of microvascular blood flow — Microvascular blood flow will be measured using a contrast enhanced ultrasound scan.
  Other Names: CEUS; Contrast enhanced ultrasound scan; SonoVue.
Other: Administration of gelofusine — Volunteers administered gelofusine in 250ml boluses
  Groups: Volunteers receiving gelofusine

SUMMARY:
Although major surgery is often required to treat abdominal problems, there is a significant risk of death or complication following these operations. By using ultrasound the amount and timing of fluid patients receive during operations can be optimised and the risk of surgery reduced. However, little is known about the exact changes in blood flow in the small vessels of the body in response to fluid. A greater understanding of this may allow for more appropriate care of patients undergoing this type of surgery in the future.

In this study of healthy volunteers we will attempt to better understand how fluid administration guided by ultrasound effects blood flow in large and small vessels, by using two different techniques of ultrasound imaging. A narrow bore (approximately 4-5mm diameter) ultrasound probe will be passed through the nostril and mouth to rest within the oesophagus allowing measurement of blood flow in the main artery, while a second probe will be rested on the volunteer's abdomen and used to record changes in blood flow in small liver blood vessels. Comparison of these two techniques during the administration of fluid will allow us to better understand the relationship between large and small vessel blood flow.

Because different types of fluid may behave in different ways, we will test the effect of two types of fluid commonly used in clinical practice; 'normal' saline solution and gelofusine.

DETAILED DESCRIPTION:
Optimizing intravascular volume and cardiac output are essential to ensure adequate organ perfusion in patients who are undergoing major surgery. To enable this cardiac output is frequently monitored during operation using a variety of techniques; one such technique is trans-oesophageal Doppler ultrasound also known as oesophageal Doppler monitoring (ODM). ODM measurement of cardiac output is a less invasive technique than many currently used methods, and has recently been recommended by NICE for adoption in clinical practice.

The matching of microvascular blood flow, cardiac output and fluid administration is advantageous for visceral organs, in marrying demands for oxygen and nutrients to their delivery. However, although there is evidence to suggest that intraoperative ODM directed fluid administration can improve outcomes in the perioperative period, reducing hospital stay and complications, there is little direct evidence that optimization of cardiac output via ODM improves the microvascular blood flow to the visceral organs which are frequently compromised by major surgical interventions. A greater appreciation of the effect of ODM guided fluid replacement on the delivery of blood and hence oxygen and nutrients to these vital organs could help with the development of more refined algorithms for fluid administration in a clinical setting in the future. In our clinical physiology laboratories we regularly employ contrast-enhanced ultrasound (CEUS) using a Phillips iU22, to visualize microvascular blood flow in healthy young and elderly men following a variety of physiological challenges. This minimally invasive ultrasound based imaging technique is ideal for gaining an insight into the effect various physiological interventions have on tissue blood flow and could be readily used to chart changes in visceral microvascular flow following ODM guided fluid optimization. Transference of this investigative approach to a clinical setting has the potential to greatly improve the care of the surgical patient requiring fluid resuscitation.

Different types of intravenous fluids are used in clinical practice. These are primarily crystalloid solutions, such as 0.9% sodium chloride ('normal' saline), or colloidal suspensions, such as gelofusine. There is good experimental evidence that the colloid gelofusine produces a greater effect on cardiac output than an equivalent volume of of saline, but it is unclear if this effect is replicated in the microvasculature.

We will test the hypotheses: (1) cardiac output and stroke volume as measured by ODM are determinants of visceral microvascular blood flow (2) visceral microvascular blood flow in elderly individuals is more closely determined by stroke volume (3) gelofusine produces a greater increase in microvascular blood flow than the same volume of normal saline.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18-80 years
* body mass index 20-30kg/m2

Exclusion Criteria:

* BMI < 20 or > 30 kg/m2.
* Active cardiovascular disease: uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arhythmias , right to left cardiac shunt or recent cardiac event.
* Individuals taking beta-adrenergic blocking agents.
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)..
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes.
* Active inflammatory bowel disease, or renal disease,
* Malignancy
* Clotting dysfunction
* Previous oesophageal surgery
* Individuals with a known history of oesophageal varices
* Individuals with a known history of epistaxis
* Family history of early (<55y) death from cardiovascular disease.
* Known sensitivity to SonoVue
* Known sensitivity to gelofusine

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male volunteers, aged 18-80.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in microvascular visceral blood flow | 30 minutes
  Microvascular visceral blood flow is assessed using contrast enhanced ultrasound scanning, following stroke volume optimisation.

SECONDARY OUTCOMES:
Change in stroke volume | 30 minutes
  The change in stroke volume will be assessed using an Oesophageal Doppler Monitor, and will be assessed pre- and post-intravenous fluid administration.
Change in haematocrit | 60 minutes
  The change in the haematocrit will be measured pre- and post-intravenous fluid administration.

CONTACTS AND LOCATIONS:
Overall Officials: John P Williams, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, School of Medicine, Division of Medical Sciences and Graduate Entry Medicine, Derby, Derbyshire, United Kingdom